CLINICAL TRIAL: NCT03187457
Title: PreFem: "What Happens to the Vaginal Microbiota When a BV Infection is Treated With Metronidazole?"
Acronym: PreFem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danisco (Industry)
Collaborators: Community Pharmacology Services Ltd (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NH-03708
Record Dates: First submitted 2017-05-18; First posted 2017-06-15 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Other): Metronidazole 400 mg 3 times daily for 5 days for Bacterial Vaginosis (BV) infection
  Interventions: Other: Metronidazole
- Control group (Other): Healthy women without Bacterial Vaginosis and without treatment
  Interventions: Other: Control: no treatment

INTERVENTIONS:
Other: Metronidazole — Women with Bacterial Vaginosis treated with Metronidazole for 5 days
  Arms: Treatment group
Other: Control: no treatment — Healthy women without Bacterial Vaginosis
  Arms: Control group

SUMMARY:
The study will assess vaginal microbiota levels before and after antibiotic treatment in females infected with Bacterial Vaginosis (BV).

DETAILED DESCRIPTION:
This method validation study will endeavour to obtain evidence for:

* Recruitment methodology effectiveness
* The usefulness of the "Canestest" test as a screening tool
* The time required for the vaginal microbiota (particularly Lactobacillus count) to return to normal after treatment of BV infection with metronidazole.
* The time required for the Nugent Score to return to normal after treatment of BV infection with metronidazole.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Female gender
* Over 18 years of age
* Have a high probability for compliance with and completion of the study

Exclusion Criteria:

* Hypersensitivity to metronidazole --only applies to Group 2.
* Post-menopausal defined as at least 12 consecutive months without menstruation
* Treatment of BV in last 4 weeks
* Clinically significant menstrual irregularities
* Suspected presence of STDs or other vaginal infection
* Pregnancy
* Breast feeding
* Participation in other clinical studies which could influence genitourinary tract microbiota
* Substance abuse
* Investigator believes that the participant may be uncooperative and/or noncompliant and should therefore not participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Change in vaginal microbiota assessed with sequencing | Baseline, at day 8, and at day 15
  Change in vaginal microbiota is assessed with sequencing at 3 time points (baseline, at day 8 and at day 15 time points post antibiotic treatment.)

SECONDARY OUTCOMES:
Vaginal microbiota/lactobacilli levels with Nugent scoring | Baseline, at day 8, and at day 15
  Nugent scoring is used for the evaluation of the vaginal microbiota at baseline, at 8 and 15 day time points post antibiotic treatment.
Diagnosis of BV with "Canestest" | Baseline
  "Canestest" will be used to diagnose BV infection at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Crawford, MD, Principal Investigator — CPS Research
Locations (1):
- CPS Research, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD